CLINICAL TRIAL: NCT06314555
Title: Impact of the sFlt-1/PlGF Ratio on Medical Decision-making and on Maternal and Neonatal Outcomes in Women Suspected of Preeclampsia
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: CEROG2023
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Preeclampsia Possible
Keywords: Preeclampsia; Soluble fms-like tyrosine kinase; Placental growth factor; Medical care decision; Hospitalization
MeSH Terms: conditions — Pre-Eclampsia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women under 37 weeks of gestation age: A woman with suspected preeclampsia and with inclusion criteria receives a blood sample, according to the department's usual practices, to analyse the values of sFlt-1 and PlGF and the usual vascular-renal sample. The woman gave her verbal consent to participate in the study. The Roche Elecsys® immunoassay sFlt-1/PlGF ratio was used to measure the two markers in the patients' blood.
  Interventions: Other: Blood sample; Other: Vascular-renal sample
- Women above 37 weeks of gestation age: A woman with suspected preeclampsia and with inclusion criteria receives a blood sample, according to the department's usual practices, to analyse the values of sFlt-1 and PlGF and the usual vascular-renal sample. The woman gave her verbal consent to participate in the study. The Roche Elecsys® immunoassay sFlt-1/PlGF ratio was used to measure the two markers in the patients' blood.
  Interventions: Other: Blood sample; Other: Vascular-renal sample

INTERVENTIONS:
Other: Blood sample — Blood sample to analyse the values of sFlt-1 and PlGF
Other: Vascular-renal sample — Usual vascular-renal sample to analyse the values of sFlt-1 and PlGF

SUMMARY:
Previous studies demonstrated that Placental Growth Factor (PIGF) and Vascular Endothelial Growth Factor (VEGF) produced by trophoblast cells decreases during Preeclampsia, whereas soluble fms-like tyrosine kinase-1 (sFlt-1), an antiangiogenic factor, increases. The ratio sFlt-1/PlGF has a higher positive predictive value than the isolated measurement. A ratio under 38 exclude risk of imminent preeclampsia and allows to outpatient follow-up with a negative predictive value of 99.3%. A ratio equal or higher than 38 permits to direct high-risk patients towards hospitalization with a positive predictive value of 36.7% of preeclampsia at 4 weeks. These findings suggest that the ratio can be used to select more appropriately women needing hospitalization for suspected preeclampsia.

DETAILED DESCRIPTION:
This is a single-center prospective and observational study conducted from the 1rst of October 2019 to the 27th of January 2021, including pregnant women suspected of preeclampsia, above 24 weeks of gestation. Values were measured using the Elecsys sFlt-1/PlGF immunoassay ratio. The investigators observed the clinical decision regarding hospitalization, intensive patient monitoring, corticosteroid administration, and labor induction before and after knowing the ratio value.

ELIGIBILITY:
Inclusion Criteria:

* pregnant patients over 24 weeks of amenorrhea
* aged 18 and over
* with suspicion of preeclampsia defined by the appearance of pregnancy-induced hypertension (≥ 140 in systolic and/or 90 mmHg in diastolic pressure over 2 measurements at 4 hours intervals) OR proteinuria (≥ 0.3 g per 24 hours).
* who systematically gave oral consent after submitting the information sheet

Exclusion Criteria:

* pregnant women with both hypertension and proteinuria because they already have a confirmed diagnosis of preeclampsia.
* receiving antihypertensive treatment before pregnancy
* or refusing to participate in the study The sFlt-1/PlGF ratio was measured only when clinically indicated as per the investigator's judgment.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Pregnant women suspected of preeclampsia, above 24 weeks of gestation.
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Doctor's medical care decisions on Hospitalization | Day 1
  Initial medical decision (hospitalization or no) was taken before knowing the test result. Revision of the medical decision occurred when the investigators had knowledge of the sFlt-1/PlGF result.

SECONDARY OUTCOMES:
Intensive monitoring | Day 1
  Intensive monitoring decision was taken before knowing the test result. Revision of the medical decision occurred when the investigators had knowledge of the sFlt-1/PlGF result.
Corticosteroid administration for lung maturation | Day 1
  Corticosteroid administration for lung maturation decision was taken before knowing the test result. Revision of the medical decision occurred when the investigators had knowledge of the sFlt-1/PlGF result.
Birth induction | Day 1
  Birth induction decision was taken before knowing the test result. Revision of the medical decision occurred when the investigators had knowledge of the sFlt-1/PlGF result.

CONTACTS AND LOCATIONS:
Overall Officials: Tiphaine BARJAT, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No